CLINICAL TRIAL: NCT03418597
Title: Randomized, Monocentric, Controlled, Superiority Phase II Trial Evaluating Clinical Hypnosis Using Virtural Reality vs Standard Pain Management Procedure During a Musculoskelettal Biopsy
Brief Title: Trial Evaluating Hypnosis Using Virtural Reality vs Standard Pain Management During Musculoskelettal Biopsy
Acronym: REVENRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET17-066 (REVENRI)
Record Dates: First submitted 2018-01-05; First posted 2018-02-01 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Musculoskeletal Cancers
Keywords: Virtual reality; Radio-guided biopsy; Pain; Anxiety; Patient's satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep local anesthesia + Virtual reality (Experimental): Pre-medication procedures and lidocaïne injection are the same as in the current practice. During the intervention delay, the patient will also experience hypnosis through a virtual reality procedure .
  Interventions: Procedure: Deep local anesthesia + Virtual reality
- Deep local anesthesia alone (Active Comparator): The musculoskeletal biopsy is performed according to the standard practice using a deep local anesthesia with premedication and lidocaïne.
  Interventions: Procedure: Deep local anesthesia alone

INTERVENTIONS:
Procedure: Deep local anesthesia + Virtual reality — Biopsy performed according to current practice (deep local anesthesia with premedication and lidocaïne). Patient will have a 3-D immersive experience, created using a visual and audio headset and a software labelled as medical device.
  Arms: Deep local anesthesia + Virtual reality
Procedure: Deep local anesthesia alone — Biopsy performed according to current practice (deep local anesthesia with premedication and lidocaïne).
  Arms: Deep local anesthesia alone

SUMMARY:
The primary objective of this trial is to evaluate the benefit of the virtual reality technology in the pain management for patients having a radio-guided musculoskeletal biopsy indication

DETAILED DESCRIPTION:
During the last years, the percutaneous biopsies took a growing importance in the diagnosis of musculoskeletal cancers. The most important advantages of percutaneous biopsies are: 1) Often performed under local anesthesia in out-patient department, 2) No visible scars, 3) Surgical intervention avoided in case of benign tumor with a low level of complications (infection, hematoma, pain).

The technology improvement of percutaneous biopsy leads to a high diagnosis success rate (80.8% for bone tumors and 83.2% for soft tissues tumors') with a low complication rate (0.7%) and then justifies the use of percutaneous biopsy as first-line diagnostic exam.

During a percutaneous biopsy, the pain is frequently felt with an increase in the "pain numeric scale" evaluated after the procedure.

The nitrous oxide is a gas mixture which can be used for its anesthetic and antalgic properties, making the pain tolerable for the patients during short procedures. However, it can cause adverse events such as nausea, vomiting and nervous system affections (excessive sedation, anxiety). Moreover, this gas is not always efficient for the pain management.

Other options have been investigated such as hypnosis and music therapy which improve patients' experience of the medical interventional procedures.

The virtual reality is a digital tool existing for about 10 years. It enables to isolate a patient from the real world which can be useful in some medical indications. It is a 3-D immersive experience, created using a visual and audio headset. Virtual reality can reduce the pain experienced during surgical interventions and has widely shown its interest in algogenic cares.

While the results are promising, a recent review of the literature shows that very few randomized clinical trials document the virtual reality benefit in pain and/or anxiety management for burn patients or patients suffering from acute or chronic pains.

The objective of this study is to demonstrate the benefit of the virtual reality in addition to a deep local anesthesia vs a deep local anesthesia alone in the pain management linked to musculoskeletal tumors biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged >= 18 years at the day of consenting to the study (no upper limit)
* Requiring a radio-guided biopsy of the musculoskeletal system,
* Informed and signed consent,
* Patient covered by a medical insurance.

Exclusion Criteria:

* Deaf patient;
* Visually-impaired patient;
* Claustrophobic and/or aquaphobic patient;
* Contraindication to a musculoskeletal biopsy, including to the premedication protocol and to the lidocaine;
* Person deprived of liberty or placed under guardianship;
* Absence of French language skills;
* History of psychiatric disease such as paranoia, schizophrenia, manic-depressive psychosis, patient with a high risk of suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Evaluate the benefit of the virtual reality in the pain management of patients needing a radio-guided musculoskeletal biopsy. | Day 0
  The main outcome will be the pain level auto-evaluated by the patient using a numeric scale composed of 11 graduations (from 0 to 10)

SECONDARY OUTCOMES:
Evaluate in both arms, the pain linked to the biopsy procedure using a numeric scale graduated from 0 to 10. | Day 1 (+/-2h) post biopsy
  The score " 0 " corresponds to " No pain " and the score " 10 " corresponds to " Maximum amount of imaginable pain "
Evaluate in both arms, the anxiety linked to the biopsy procedure using a numeric scale graduated from 0 to 10 | Day 0
  The score " 0 " corresponds to " No anxiety " and the score " 10 " corresponds to " Maximum imaginable anxiety "
Evaluate the analgesics consumption in both arms | through study completion, an average of 24 hours
  Evaluation according to the following classification and recording the dosages and units taken: Level 1 - Non morphinic analgesics; Level 2 - Weak opioides analgesics; Level 3 - Strong opioides analgesic
Evaluate the global satisfaction of patients in both arms | Day 0
  The score "0" corresponds to " Absence of satisfaction " and the score " 10 " corresponds to " Full satisfaction ".
Evaluate costs in both arms | through study completion, an average of 24 hours
  Evaluation of costs involved for the patient's treatment and care

CONTACTS AND LOCATIONS:
Overall Officials: BOUHAMAMA Amine, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France